CLINICAL TRIAL: NCT00365781
Title: A Phase 1, Open-Label Examination of the Dermatologic Effects From Subcutaneous Administration of ISIS 113715, and Antisense Oligonucleotide Inhibitor of Protein Tyrosine Phosphatase 1B, in Healthy Volunteers
Brief Title: Examination of Dermatologic Effects From Subcutaneous Injections of ISIS 113715
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 113715-CS13
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2007-10-17 (Estimated); Status verified 2007-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Injection Site Reaction; Subcutaneous administration; Dermatological effects; Antisense
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Injection Site Reaction | interventions — ISIS-113715

INTERVENTIONS:
Drug: ISIS 113715

SUMMARY:
10 healthy volunteers will be enrolled to each receive two subcutaneous injections of ISIS 113715 in the abdomen on Study Day 1. Each subject will receive their two injections within a 5-minute period. On Study Days 2 and 8, each subject's injection sites will be assessed for dermatologic effects. The Isis Project Physician(s) will observe the injection sites on Study Day 2 and may also observe on Study Day 8.

Routine clinical chemistry, hematology, and urinalysis tests will be performed on Study Day 1 and Day 8. Subjects will be contacted by telephone on Study Day 30 to monitor for the occurrence of new serious adverse events (SAEs). Thereafter, the subjects will be discharged from the study.

DETAILED DESCRIPTION:
Following a two-week period for subject screening, 10 eligible subjects will be dosed subcutaneously with ISIS 113715 on a single calendar date (Study Day 1). Each subject will receive two subcutaneous injections given within a 5-minute period. The first injection will be 200 mg ISIS 113715 given in 1.0 mL and will be injected about 7.5 cm to the left of the umbilicus. The second injection will be 200 mg ISIS 113715 given in 2.0 mL and will be injected about 7.5 cm to the right of the umbilicus. Both injections will be delivered using 3.0-mL syringes outfitted with 30-gauge, 0.5-inch needles. To further minimize variability, all injections will be performed by a single individual, the Investigator or his designee, employing uniform technique for all of the injections.

Dermatologic responses at injection sites will be assessed at 1 and 7 days after the injections (Study Days 2 and 8, respectively). Effects will be evaluated through completion of the Injection Site Assessment Questionnaires by the Investigator and the recording of adverse events reported by the subject or observed by the Investigator. The Isis Project Physician(s) will observe the injection sites on Study Day 2 and may also observe on Study Day 8.

Routine clinical chemistry, hematology, and urinalysis tests will be performed on Study Days 1 (prior to administration of ISIS 113715) and 8.

Subjects will be contacted by telephone on Study Day 30 to monitor for the occurrence of new serious adverse events. Thereafter, the subjects will be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female: Females are post menopausal or surgically sterile; Males are surgically sterile, abstinent, or utilizing an acceptable barrier contraceptive method. Must also agree to continue abstinence and/or to use an acceptable barrier contraceptive method for at least four weeks after their injections of ISIS 113715
* Aged 18 to 65 years
* Weight > 50 kg
* Body mass index > 29 kg/m²

Exclusion Criteria:

* Pregnant, breastfeeding, or intends to become pregnant
* Positive hepatitis B virus, hepatitis C virus, or HIV test
* History of clinical significant abnormalities in complement or coagulation parameters or taking medication that may affect coagulation (e.g., heparin, warfarin), except aspirin or non-steroidal anti-inflammatory agents (NSAID)
* Current or history of significant skin disorders
* History of alcohol or drug abuse
* History of liver or renal disease
* Malignancy (with the exception of basal or squamous cell carcinoma of the skin if adequately treated and no recurrence for > one year)
* Liver function tests greater than the Upper Limit of Normal (ULN)
* Clinically significant and currently active diseases or active infection requiring antiviral or antimicrobial therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-08; Study Completion 2006-09

PRIMARY OUTCOMES:
Compare the dermatologic responses to 200 mg/1.0 mL and 200 mg/2.0 mL ISIS 113715 administered subcutaneously into separate abdominal sites, with both injections given on the same day.
Evaluate and examine the effect of treatment on laboratory results, vital signs, and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Wedel, MD, JD, FACP, Study Director — Ionis Pharmaceuticals, Inc.
Locations (1):
- Therapeutics Clinical Research, San Diego, California, United States